CLINICAL TRIAL: NCT05853367
Title: A Phase 1/1b Open-label, Multicenter Clinical Study of MK-0472 as Monotherapy and Combination Therapy in Participants With Advanced/Metastatic Solid Tumors.
Brief Title: Study of MK-0472 in Participants With Advanced/Metastatic Solid Tumors (MK-0472-001)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0472-001; MK-0472-001 (Other: MSD); 2024-516006-32-00 (Registry Identifier: EU CT); U1111-1310-1179 (Registry Identifier: UTN)
Record Dates: First submitted 2023-05-02; First posted 2023-05-10 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Solid Tumors; Advanced Solid Tumors
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Death-Ligand 1 (PDL1, PD-L1); Src Homology-2 Domain Containing Protein Tyrosine Phosphatase-2 (SHP-2)
MeSH Terms: conditions — Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- MK-0472 (Experimental): Participants receive MK-0472 via oral capsule according to one of the protocol-specified dosing regimens until disease progression or withdrawal/discontinuation.
  Interventions: Drug: MK-0472
- MK-0472 + Pembrolizumab (Experimental): Participants receive MK-0472 via oral capsule according to one of the protocol-specified dosing regimens until disease progression or withdrawal/discontinuation, plus pembrolizumab 200 mg via intravenous (IV) infusion on Day 1 of each 3-week cycle for up to 35 cycles (up to approximately 2 years).
  Interventions: Drug: MK-0472; Biological: Pembrolizumab
- MK-0472 + MK-1084 (Experimental): Participants receive MK-0472 via oral capsule according to one of the protocol-specified dosing regimens, plus MK-1084 via oral capsule until disease progression or withdrawal/discontinuation.
  Interventions: Drug: MK-0472; Drug: MK-1084

INTERVENTIONS:
Drug: MK-0472 — Oral Administration
Biological: Pembrolizumab — IV infusion
  Other Names: MK-3475; Keytruda®
  Arms: MK-0472 + Pembrolizumab
Drug: MK-1084 — Oral Administration
  Arms: MK-0472 + MK-1084

SUMMARY:
The purpose of this study is to assess the efficacy, safety, and tolerability of MK-0472 administered as monotherapy and in combination with pembrolizumab (MK-3475) or MK-1084 in participants with histologically or cytologically confirmed diagnosis of advanced/metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Has histologically or cytologically confirmed solid tumor by pathology report that is advanced/metastatic
* Participants who are hepatitis B surface antigen (HBsAg) positive are eligible if they have received HBV antiviral therapy for at least 4 weeks, and have undetectable HBV viral load prior to study enrollment
* Participants with history of hepatitis C virus (HCV) infection are eligible if HCV viral load is undetectable at screening
* Participants with human immunodeficiency virus (HIV) infection must have well controlled HIV on stable (>4 weeks) antiretroviral therapy (ART)
* Arm 1: Oncogenic receptor tyrosine kinase (RTK) pathway alterations confirmed by a historical report or local testing (tissue or blood) and have received, or been intolerant to, all available treatment known to confer clinical benefit
* Arm 2: Tumor types known to be sensitive to anti-programmed cell death 1 protein (PD-1)/ligand 1 (L1) therapies are eligible. Tumor types permitted include: melanoma, non-small cell lung cancer (NSCLC) without epidermal growth factor receptor (EGFR)/anaplastic lymphoma kinase (ALK)/ROS1 mutations, renal cell carcinoma, urothelial carcinoma, Merkel cell carcinoma, MSI-high CRC, endometrial cancer, cervical cancer, small cell lung cancer, triple negative breast cancer, esophageal cancer, gastric cancer, biliary tract cancer, hepatocellular carcinoma, head and neck squamous cancer, cutaneous squamous cancer, anal squamous cancer, and mesothelioma
* Arm 3: Has histologically OR blood-based confirmation of Kirsten rat sarcoma viral oncogene homolog (KRAS) G12C mutation

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* Has not recovered to common terminology criteria for adverse events (CTCAE) Grade 1 or better from any adverse events that were due to cancer therapeutics administered more than 4 weeks earlier. Participants receiving ongoing replacement hormone therapy for endocrine immune-related AEs will not be excluded from participation in this study
* Has history of a second malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 2 years
* History of hyperparathyroidism or hypercalcemia
* Has one or more of the following ophthalmological findings/conditions: a) Intraocular pressure >21 mm Hg and/or any diagnosis of glaucoma b) Diagnosis of central serous retinopathy, retinal vein occlusion, or retinal artery occlusion and c) Diagnosis of retinal degenerative disease
* Has clinically significant cardiovascular disease
* Bullous exfoliative skin disorders of any grade
* Known hypersensitivity to MK-0472, MK-1084, or pembrolizumab, or any of their excipients
* Received therapy with a proton-pump inhibitor or an H2 histamine blocker receptor antagonist within 7 days before the first scheduled day of study dosing
* Has discontinued prior therapy with an anti-programmed cell death-1 (PD-1), anti-programmed death-ligand 1 (PD-L1), or anti-programmed death-ligand 2 (PD-L2) agent or with an agent directed to another stimulatory or coinhibitory T-cell receptor due to an adverse event
* Received prior systemic anticancer therapy including investigational agents within 4 weeks before first dose
* Received a live or live-attenuated vaccine within 30 days before the first dose of study intervention
* Has received an investigational agent or has used an investigational device within 4 weeks prior to study intervention administration
* Has diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study medication
* Has known additional malignancy that is progressing or has required active treatment within the past 2 years
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable for at least 4 weeks as confirmed by repeat imaging performed during the study screening, are clinically stable and have not required steroid treatment for at least 14 days before the first dose of study intervention
* Has active autoimmune disease that has required systemic treatment in the past 2 years except replacement therapy
* Has history of pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease
* Has active infection requiring systemic therapy
* Has history of allogeneic tissue/solid organ transplant
* Have not adequately recovered from major surgery or have ongoing surgical complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2023-07-06 (Actual); Primary Completion 2028-02-12 (Estimated); Study Completion 2028-02-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Who Experience a Dose Limiting Toxicity (DLT) as Assessed Using Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 | At the end of Cycle 1 (each cycle is 21 days)
  DLT will be defined as any drug-related AE observed during the DLT evaluation period (e.g. Cycle 1) that results in a change to a given dose or a delay in initiating the next cycle.
Number of Participants Who Experience One or More Adverse Events (AEs) | Up to approximately 56 months
  An AE is defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment. The number of participants who experience one or more AE's will be reported.
Number of Participants Who Discontinue Study Treatment Due to an Adverse Event (AE) | Up to approximately 56 months
  An AE is defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment. The number of participants who discontinue study treatment due to an AE will be reported.

SECONDARY OUTCOMES:
Area Under the Concentration Time-curve From Time 0 to the End of the Dosing Period (AUCtau) of MK-0472 | At predetermined timepoints predose and postdose up to Cycle 6 (Each cycle length = 21 Days)
  Blood samples will be collected at specified intervals for the determination of AUCtau. AUCtau is defined as the area under concentration-time curve from 0 to the end of the dosing period.
Lowest Plasma Concentration (Ctrough) of MK-0472 | At predetermined timepoints Predose up to Cycle 6 (Each cycle length = 21 Days)
  Blood samples will be collected at specified intervals for the determination of Ctrough. Ctrough is defined as the lowest concentration of MK-0472 reached before the next dose is administered.
Maximum Plasma Concentration (Cmax) of MK-0472 | At predetermined timepoints postdose up to Cycle 6 (Each cycle length = 21 Days)
  Blood samples will be collected at specified intervals for the determination of Cmax. Cmax is defined as the maximum concentration of MK-0472 reached.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (25):
- United States (4):
  - Northwestern Memorial Hospital ( Site 0002), Chicago, Illinois
  - The University of Louisville, James Graham Brown Cancer Center ( Site 0004), Louisville, Kentucky
  - John Theurer Cancer Center at Hackensack University Medical Center ( Site 0001), Hackensack, New Jersey
  - Rutgers Cancer Institute of New Jersey ( Site 0005), New Brunswick, New Jersey
- Canada (3):
  - Princess Margaret Cancer Centre ( Site 0101), Toronto, Ontario
  - Centre Hospitalier de l'Université de Montréal-Unit for Innovative Therapies ( Site 0100), Montreal, Quebec
  - Jewish General Hospital ( Site 0104), Montreal, Quebec
- Chile (4):
  - Centro de Estudios Clínicos SAGA ( Site 0701), Santiago, Region M. de Santiago
  - Fundacion Arturo Lopez Perez ( Site 0700), Santiago, Region M. de Santiago
  - Centro de Investigacion Clinicadela Universidad Catolica ( Site 0703), Santiago, Region M. de Santiago
  - Bradfordhill ( Site 0702), Santiago, Region M. de Santiago
- Israel (5):
  - Rambam Health Care Campus ( Site 0304), Haifa
  - Shaare Zedek Medical Center ( Site 0303), Jerusalem
  - Rabin Medical Center ( Site 0301), Petah Tikva
  - Sheba Medical Center ( Site 0300), Ramat Gan
  - Sourasky Medical Center ( Site 0302), Tel Aviv
- Poland (2):
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - Panstwowy Instytut Badawczy w Warszawie ( Site 0401), Warsaw, Masovian Voivodeship
  - Uniwersyteckie Centrum Kliniczne ( Site 0400), Gdansk, Pomeranian Voivodeship
- Spain (4):
  - Institut Català d'Oncologia - L'Hospitalet-Medical Oncology ( Site 0501), L'Hospitalet de Llobregat, Catalonia
  - Centro Integral Oncologico Clara Campal-Hospital HM Universitario Sanchinarro-START Madrid, ( Site 0504), Madrid, Madrid, Comunidad de
  - Hospital Universitari Vall d'Hebron ( Site 0500), Barcelona
  - Hospital Virgen del Rocio ( Site 0503), Seville
- Switzerland (3):
  - Hôpitaux Universitaires de Genève (HUG) ( Site 0202), Geneva, Canton of Geneva
  - Cantonal Hospital St.Gallen-Oncology & Hematology ( Site 0201), Sankt Gallen, Canton of St. Gallen
  - Ospedale Regionale Bellinzona e Valli ( Site 0200), Bellinzona, Canton Ticino

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26116&tenant=MT_MSD_9011